CLINICAL TRIAL: NCT06827951
Title: A Mixed-Methods Approach Utilizing Self-Report Scales and Oxytocin Levels to Determine the Potential Benefits of Parent Child Interaction Therapy (PCIT)
Brief Title: Potential Benefits of Parent Child Interaction Therapy (PCIT)
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202400867
Record Dates: First submitted 2024-11-18; First posted 2025-02-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Autonomic Dysregulation; Anxiety; Depression; Parent-Child Relations
Keywords: Polyvagal Theory; Adversity; Parent-Child Interaction Therapy; Attachment; Autonomic Reactivity; Oxytocin
MeSH Terms: conditions — Primary Dysautonomias; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Saliva samples will be collected at two timepoints (pre PCIT and during PCIT). Salivary samples will be used to measure oxytocin levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCIT Group: All participants will complete the five online surveys and provide two saliva samples.
  Interventions: Behavioral: Parent-Child Interaction Therapy (PCIT)

INTERVENTIONS:
Behavioral: Parent-Child Interaction Therapy (PCIT) — Participants will undergo the standard PCIT program, which consists of two phases: Child-Directed Interaction (CDI) and Parent-Directed Interaction (PDI).
  * CDI Phase: Parents will learn and practice techniques that focus on strengthening the parent-child relationship through play and positive reinforcement.
  * PDI Phase: Parents will be coached in effective discipline strategies to manage their child's behavioral problems.

SUMMARY:
The goal of this study is to explore possible benefits of Parent-Child Interaction Therapy (PCIT). The main goals of the study are:

* To investigate whether pre-survey measures of autonomic reactivity relate to the overall functioning of participants.
* To examine the effects of PCIT To identify individual characteristics that influence the effects of PCIT.

Participants will:

* complete 5 online surveys (1x pre-PCIT, 3x during PCIT, and 1x post-PCIT)
* complete the PCIT program

DETAILED DESCRIPTION:
It is the specific intent of this proposal to experimentally explore the possible benefits and mechanisms through which PCIT can influence self-reported stress and autonomic and neuroendocrine functioning in parents. This will be accomplished by our team by using well-validated self-report measures of mental health, autonomic reactivity, parental stress and attachment, and non-invasive measurements of levels of oxytocin.

Specific Aim 1: To investigate whether pre-intervention measures of ANS reactivity and the neuropeptides oxytocin relate to the overall functioning of the participants.

* The investigators will examine how measures of autonomic reactivity and levels of oxytocin relate to prior mental/medical health.
* Hypothesis: Participants with lower levels of oxytocin and/or increased autonomic reactivity will report being more impacted by their prior adversity and having more emotional/physical symptoms.

Specific Aim 2: To investigate the impact of PCIT

* The investigators will explore whether PCIT leads to improvements in parental stress, parent-child attachment, and parental neuroendocrine functioning.
* Hypothesis: Parents will show a significant decrease in perceived stress and improvement in emotional wellbeing oxytocin levels following CDI. They will also show a decrease in perceived stress, and improvement in attachment and emotional wellbeing following the entire PCIT intervention.

Specific Aim 3: To identify individual characteristics that influence the effectiveness of PCIT.

* The investigators will explore the impact of specific vulnerability and resiliency factors (e.g., stress, prior adversity) on how well parents benefit from PCIT
* Hypothesis: Parental stress and prior mental/medical adversity will negatively impact the effectiveness of intervention

ELIGIBILITY:
Inclusion Criteria:

* Parents of children aged 2-7 years old who are eligible for Parent-Child Interaction Therapy (PCIT) based on behavioral concerns.
* The primary caregiver of the child and be actively involved in the child's daily care.
* Willing to attend all PCIT sessions and complete pre-, mid- and post-intervention assessments.
* Fluent in English to ensure comprehension of the intervention and assessment materials.

Exclusion Criteria:

* Parents with diagnosed severe mental health disorders (e.g., schizophrenia, bipolar disorder) that may interfere with participation in PCIT.
* Children with conditions that require interventions other than PCIT (e.g., severe developmental disabilities).
* Parents who have previously participated in PCIT are excluded to avoid confounding results.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators intend to recruit parents of children aged 2-7 with behavioral issues who are eligible for the PCIT program at two university clinics (UF Health Jacksonville and Shands Gainesville) specializing in child psychology and parent training. This population represents those most likely to experience stress and benefit from improved parent-child interactions and stress regulation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Measuring Change in Autonomic Reactivity using the Body Perceptions Inventory Short Form | Through study completion, an average of 20 weeks
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Assessing the Impact of Adversity History | Up to 1 week
  This measure assesses the impact of six types of traumatic experiences (childhood adverse experiences, childhood maltreatment, intimate partner maltreatment, other person maltreatment, life-threatening situations, sudden losses, and person health situations). Each item is scored on a 5-point Likert scale (did not occur = 0, occurred and no impact on my life = 1 to big impact on my life = 4). Items are summed to determine total impact scores.
Measuring change in oxytocin Levels | Up to 4 weeks
  Oxytocin levels will be assessed using salivary samples. Increased salivary oxytocin indicates improvement.
Measuring change in parental stress using the parental stress scale | Through study completion, an average of 20 weeks
  This 18-item questionnaire assesses parents' feelings about their parenting role via a 5-point Likert scale (Strongly disagree = 1 to Strongly agree = 5). Lower scores indicate lower levels of parental stress.
Measuring change in parental attachment using the Child-Parent Relationship Scale | Through study completion, an average of 20 weeks
  This 30-item questionnaire assesses parents' views of their relationship with their child via a 5-point Likert scale (1 = definitely does not apply to 5 = definitively applies). The scores for the subscales (e.g., closeness, conflict, dependency) are calculated by summing the relevant items, with higher scores indicating more positive views of the relationship.
Measuring change in child behavior using the parent-report Eyberg Child Behavior Inventory | Through study completion, an average of 20 weeks
  This 36-item measure assesses the frequency and severity of disruptive behaviors, as well as the extent to which parents find the behaviors troublesome via a 7-point Likert scale (1 Never Occurs to 7 = Always Occurs) and a binary Problem scale. Total Intensity Scale scores range from 36 to 352, with clinical cut-off scores of 131-133.
Measuring change in anxiety using the General Anxiety Disorder-7 | Through study completion, an average of 20 weeks
  This 7-item measure assesses anxiety via a 4-point Likert scale (0 = Not at all to 3 = Nearly every day) with higher scores reflecting more symptoms of anxiety.
Measuring change in depression using the Patient Health Questionnaire-8 | Through study completion, an average of 20 weeks
  This 8-item measure assesses depression via a 4-point Likert scale (0 = Not at all to 3 = Nearly every day) with higher scores reflecting more symptoms of depression.
Measuring change in post-traumatic stress symptoms using the PTSD Checklist for DSM-5 | Up to 1 week
  This 20-item measure assesses PTSD symptoms via a 5-point Likert (0 = Not at all to 4 = Extremely) with higher scores reflecting more symptoms of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Britney N. Duner, LCSW, Principal Investigator — University of Florida College of Medicine Jacksonville; Liliana L. Acosta, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - UF Health Child Psychiatry, Gainesville, Florida
  - UF Health Psychiatry San Jose, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No